CLINICAL TRIAL: NCT01456416
Title: Pilot Study for Evaluation of Glatiramer Acetate in RRMS Patients With Comorbid Autoimmune Conditions
Brief Title: Glatiramer Acetate for Multiple Sclerosis With Autoimmune Comorbidities
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Other Study IDs: GAforMS with AutoimmuneComor
Record Dates: First submitted 2011-08-19; First posted 2011-10-20 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: RRMS; Multiple Sclerosis; Glatiramer Acetate; Autoimmune Comorbidities; Psoriasis; Autoimmune Thyroiditis; Vasculitis; Rheumatoid Arthritis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Psoriasis; Thyroiditis, Autoimmune; Vasculitis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glatiramer Acetate: GA administered SQ daily in MS patients who met all Inclusion-Exclusion Criteria and were approved by their Health Care Plans for GA treatment.

SUMMARY:
The incidence of autoimmune conditions is at least 2-3 times higher in Multiple Sclerosis population than in general population. These MS patients category response unfavorably to the Interferon. The investigators suggest that autoimmune co morbidity can serve as a biological marker predicting good response to GA.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an auto-immune neurodegenerative disease that affects more than 400,000 individuals in the United States, and 2.5 million worldwide (www.nationalmssociety.org). The main pathogenic mechanism in MS involves an inflammatory condition that damages the myelin of the central nervous system (CNS), resulting in axonal damage and neurological impairment, often leading to severe disability. MS is one of the most common causes of neurological disability in young and middle-aged adult individuals, and as such has a tremendous physical, psychological and social impact on patients' lives. MS is a complex disease diagnosed by McDonald criteria with different clinical and pathological phenotypes. Several forms of MS have been described: Relapsing-Remitting (RRMS), Secondary-Progressive MS (SPMS), Progressive-Relapsing MS (PRMS), and Primary-Progressive MS (PPMS).

Glatiramer Acetate (GA) and Beta-Interferons (β-IFNs) are well established first-line immunomodulating treatment options for relapsing remitting multiple sclerosis (RRMS) with excellent safety profiles. The mechanisms of action of GA and IFNs are different. It is well known that in general Disease-Modifying Treatments (DMTs) reduce relapse rate in more than half of the multiple sclerosis (MS) patients who receive DMT, while having little if any effect on the rest. It has been speculated that the response to beta-interferons or GA may have genetic basis. As Axtell RC et al. indicated the experimental autoimmune encephalomyeilits (EAE) in mouse caused by TH1 cells generally respond well to interferon-beta, while EAE caused by TH17 cells get worse with interferon-beta.

Autoimmune disease is an extreme situation where the autoimmune response overshoots and goes out of control. The other extreme is a degenerative disorder, where the autoimmune response is not strong enough for effective protection, and degeneration therefore continues. GA being an immunomodulator may provide both properly regulated immune suppression (in the case of autoimmune disease) and properly regulated immune activation (in the case of the neurodegenerative disease).

Autoimmune conditions cluster in families with high risk for multiple sclerosis than in general population which suggests that the disease might arise on a background of a generalized susceptibility to autoimmunity. Occurrence of psoriasis, autoimmune thyroiditis, vasculitis, rheumatoid arthritis, scleroderma, lupus are seen more commonly in MS patients. Many of these patients initially get started on beta-IFNs, and usually do not do well on them. According to Investigator's and the USC MS Comprehensive Care Center experience, autoimmune co-morbidity associated with MS can serve as a biological marker predicting good response to GA and unfavorable response to the IFNs.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite multiple sclerosis defined by McDonald Criteria.
* Between 18-60 years of age.
* Subject must able to understand and sign the IRB- approved informed consent form prior to the performance of any study-specific procedures and is willing to comply with the required scheduling and assessments of the protocol.
* Subjects who are women of childbearing potential, must have a negative serum pregnancy test at the screening visit, and must be willing to practice a reliable birth-control method.
* Subjects must have officially diagnosed and documented co-morbid, other than MS, autoimmune condition (psoriasis, vasculitis, thyroiditis or rheumatoid arthritis).
* At the time of enrollment patients were on beta IFN (Avonex, Betaseron or Rebif) treatment for at least 3 months.

Exclusion Criteria:

* Women who are either pregnant or breastfeeding, and women of child-bearing potential (defined as not surgically sterile or at least two years postmenopausal) who are not using one of the following birth control methods: tubal ligation, implantable contraception device, oral, patch, injectable or transdermal contraceptive, barrier method or sexual activity restricted to vasectomized partner.
* Any clinically significant general health conditions that may interfere with the trial participation.
* Subject has a history of drug or alcohol abuse within the past year.
* Subject had corticosteroid treatment within last 90 days.
* Subject started new medication within last 30 days.
* Subject is a participant in another research project.
* Subject has contraindications for GA treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All Subjects meeting inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Global Impression Scale (CGI-1). | Comparison of CGI-1 score pre- and post-treatment.at 6 months.
  The primary objective is to determine whether daily GA injections do not aggravate comorbid autoimmune conditions.

SECONDARY OUTCOMES:
Secondary objectives include Visual Analog Scale (VAS). | Secondary objective will be done at Baseline, Mo 3, Mo 6.
  Comparison of VAS data pre- and post-treatment (Baseline, Mo 3, Mo 6).
Secondary objectives include Expanded Disability Status Scale (EDSS) | Secondary objective will be done at Baseline, Mo 3, Mo 6.
  Comparison of EDSS score pre- and post-treatment (Baseline, Mo 3, Mo 6).
Secondary objectives include concomitant medication review. | Secondary objective will be done at Baseline, Mo 3, Mo 6.
  Comparison/review of Concomitant Medications used for co-morbid condition treatment (Baseline, Mo 3, Mo 6).

CONTACTS AND LOCATIONS:
Overall Officials: Regina Berkovich, M.D.Ph.D, Principal Investigator — LAC+USC
Locations (1):
- USC MS Comprehensive Care Center & Research Group, Los Angeles, California, United States

REFERENCES:
- [Background] 1. McDonald, W.I., et al., 2001. Recommended diagnostic criteria for multiple sclerosis: guidelines from the International Panel on the diagnosis of multiple sclerosis. Ann Neurol, 2001. 50(1): p. 121-7. 2. Axtell RC, de Jong BA, Raman C,et al. T helper type 1 and 17 cells determine efficacy of interferon beta in multiple sclerosis and experimental encephalomyelitis. Nat Med 2010; 16(4):406-412. E-pub 2010 Mar 28. 3. Howard L. Weiner, MD, Multiple Sclerosis Is an Inflammatory T-Cell-Mediated Autoimmune Disease, Arch Neurol. 2004; 61:1613-1615. 4. Teitelbaum, D., A. Meshorer, T. Hirshfeld, R. Arnon, and M. Sela. 1971. Suppression of experimental allergic encephalomyelitis by a synthetic polypeptide. Eur. J. Immunol. 1:242. 5. Ben-Nun, A., I. Mendel, R. Bakimer, M. Fridkis-Hareli, D. Teitelbaum, R. Arnon, M. Sela, and N. Kerlero de Rosbo. 1996. The autoimmune reactivity to myelin oligodendrocyte glycoprotein (MOG) in multiple sclerosis is potentially pathogenic: effect of copolymer 1 on MOG-induced disease. J. Neurol.243:S14. 6. Jonathan Kipnis and Michal Schwartz, Dual action of glatiramer acetate (Cop-1) in the treatment of CNS autoimmune and neurodegenerative disorders, Trends in Molecular Medicine, Volume 8, Issue 7, 319-323, 1 July 2002, doi:10.1016/S1471-4914(02)02373-0 7. Lisa F Barcellos, Brinda B Kamdar, Patricia P Ramsay, Cari DeLoa, Robin R Lincoln, Stacy Caillier, Silke Schmidt, Jonathan L Haines, Margaret A Pericak-Vance, Jorge R Oksenberg, Stephen L Hause, Clustering of autoimmune diseases in families with a high-risk for multiple sclerosis: a descriptive study, Lancet Neurol 2006; 5: 924-31